CLINICAL TRIAL: NCT06443801
Title: The Efficiency Of Web-Based Breastfeeding Education In Pregnancy According To The Theory Of Breastfeeding Self-Efficacy
Brief Title: Efficacy Of Web-based Breastfeeding Education
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nurdan Demirci (Other)
Responsible Party: Sponsor-Investigator, Nurdan Demirci, Prof, Marmara University
Organization: Marmara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Marmara U- elıfvlgl-001
Record Dates: First submitted 2023-10-02; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Volunteering to Participate in the Study
MeSH Terms: interventions — Pregnancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THE GROUP THAT WILL NOT TAKE WEB-BASED BREASTFEEDING EDUCATION IN PREGNANCY (No Intervention): This group will not take web-based education.
- THE GROUP THAT WİLL TAKE WEB-BASED BREASTFEEDİNG EDUCATION İN PREGNANT (Experimental): this group will take web-based education.
  Interventions: Other: THE GROUP THAT WILL TAKE WEB-BASED BREASTFEEDING EDUCATION IN PREGNANCY

INTERVENTIONS:
Other: THE GROUP THAT WILL TAKE WEB-BASED BREASTFEEDING EDUCATION IN PREGNANCY — The data of the study will be applied to both groups at the same time. No training will be given to the control group, and web-based breastfeeding training consisting of 4 modules will be given to the experimental group during their pregnancy. As data collection tools; Pregnant data collection form, Postpartum information form, IOWA infant feeding attitude scale, IMDAT scale, Edinburgh depression scale, Breastfeeding motivation scale, Insufficient milk perception scale, Breastfeeding self-efficacy scale and System usability scale will be used. Data collection tools will be applied to women at pregnancy, postpartum 7th day, PP 3rd month and PP 6th month.
  Appropriate methods will be used in the evaluation of the data. The significance level will be determined as α=0.05.
  The sample of the study consisted of 90 primiparous pregnant women, 45 of whom were in the control and 45 in the experimental group, who met the inclusion criteria.
  Arms: THE GROUP THAT WİLL TAKE WEB-BASED BREASTFEEDİNG EDUCATION İN PREGNANT

SUMMARY:
Breastfeeding is the safest and healthiest method of feeding an infant and positively affects the health of both the mother and the baby in the short and long term.

Breastfeeding self-efficacy refers to the mother's perceived ability and self-confidence to breastfeed her baby.

Studies have reported that web-based support programs increase the quality of life in individuals, are useful in symptom management, and are effective in raising awareness on the subjects intended to provide support and in gaining positive attitudes and behaviors.

Today, web-based support programs are created thanks to advances in science and technology; It has advantages such as being cheap, easily accessible, not causing any harm when done under control, providing flexibility in the participant's use of time, and accessing the training content whenever needed. Due to the pandemic process, the investigators are in and with the effect of developing technology, training is provided for the needs of individuals by using many alternative education methods such as web-based education and distance education in the field of health, as in many areas. Studies have reported that web-based support programs increase the quality of life in individuals, are useful in symptom management, and are effective in raising awareness on the subjects intended to provide support and in gaining positive attitudes and behaviors.

The study is planned to be carried out between 01.01.2023 and 31.07.2024 in the Family Health Centers affiliated with the Taşköprü District Health Directorate of Kastamonu. The study universe consists of 24-36 weeks pregnant women who come to the Family Health Centers of the Taşköprü District Health Directorate. The sample of the study consisted of 90 primiparous pregnant women, 45 of whom were in the control and 45 in the experimental group, who met the inclusion criteria.

Data collection tools will be applied to women at pregnancy, postpartum 7th day, PP in the 3rd month, and PP in the 6th month.

Appropriate methods will be used in the evaluation of the data. The significance level will be determined as α=0.05.

DETAILED DESCRIPTION:
Breastfeeding is the safest and healthiest method of feeding an infant and positively affects the health of both the mother and the baby in the short and long term. Breast milk not only meets the nutritional needs of the newborn, but also protects it from many diseases, makes a great contribution to its mental and physical development, and most importantly, it provides a unique bond between mother and baby.

According to TDHS 2018 data, the rate of exclusive breastfeeding for the first six months is 41%, and this rate decreases with age. The rate of breastfeeding for 0-1-month-old children is 59%, 2-3-month-olds 45%, and 4-5-month-olds 14%.

One of the most important factors affecting breastfeeding is the mother's perception of self-efficacy. Breastfeeding self-efficacy refers to the mother's perceived ability and self-confidence to breastfeed her baby. Perception of breastfeeding self-efficacy; It determines whether the mother will breastfeed or not, how much effort she will put into it, her thoughts on breastfeeding, and her ability to cope with the difficulties she will face during the breastfeeding process emotionally.

Considering the existence of real or potential problems with breastfeeding, breastfeeding counseling is required for every expectant mother. This counseling will ensure that expectant mothers will be prepared for all kinds of breastfeeding problems that they may experience in the postpartum period. Studies have reported that web-based support programs increase the quality of life in individuals, are useful in symptom management, and are effective in raising awareness on the subjects intended to provide support and in gaining positive attitudes and behaviors.

For successful initiation, maintenance and termination of breastfeeding, mothers should be provided with a balanced diet during pregnancy, necessary breast care, physical and mental health, and training on breastfeeding.

Today, web-based support programs created thanks to advances in science and technology; It has advantages such as being cheap, easily accessible, not causing any harm when done under control, providing flexibility in the participant's use of time, and accessing the training content whenever needed. Due to the pandemic process the investigators are in and with the effect of developing technology, trainings are provided for the needs of individuals by using many alternative education methods such as web-based education and distance education in the field of health, as in many areas. Studies have reported that web-based support programs increase the quality of life in individuals, are useful in symptom management, and are effective in raising awareness on the subjects intended to provide support and in gaining positive attitudes and behaviors.

Studies on this subject are generally studies that briefly mention breastfeeding under the title of baby care and are not long enough. For this reason, the investigators aim to provide maximum benefit by giving this training to expectant mothers who have never given birth before, that is, who will breastfeed their baby for the first time, by addressing the issue of breastfeeding only.

The study is planned to be carried out between 01.01.2023 and 31.07.2024 in the Family Health Centers affiliated to the Taşköprü District Health Directorate of Kastamonu. The universe of the study consists of 24-36 weeks pregnant women who come to the Family Health Centers of the Taşköprü District Health Directorate. The sample of the study consisted of 90 primiparous pregnant women, 45 of whom were in the control and 45 in the experimental group, who met the inclusion criteria.

The data of the study will be applied to both groups at the same time. No training will be given to the control group, and web-based breastfeeding training consisting of 4 modules will be given to the experimental group during their pregnancy. As data collection tools; Pregnant data collection form, Postpartum information form, IOWA infant feeding attitude scale, IMDAT scale, Edinburgh depression scale, Breastfeeding motivation scale, Insufficient milk perception scale, Breastfeeding self-efficacy scale and System usability scale will be used. Data collection tools will be applied to women at pregnancy, postpartum 7th day, PP 3rd month and PP 6th month.

Appropriate methods will be used in the evaluation of the data. The significance level will be determined as α=0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in the study.
2. Being primiparous at 24-36 weeks of pregnancy.
3. To be able to speak and speak Turkish.
4. To be at least a primary school graduate.
5. Having a computer or smartphone at home and being able to use it.
6. No risk in pregnancy.
7. The woman does not have any chronic disease.

Exclusion Criteria:

1. The emergence of a risky situation during pregnancy.
2. Premature birth of the woman participating in the study.
3. Carrying out a risky birth and hospitalization of the mother or baby due to it.
4. Termination of pregnancy prematurely for any reason (such as infant death)
5. The fact that the pregnant women in the experimental group did not complete the training modules before birth.
6. The fact that the women participating in the study did not respond to the directed scales and questionnaires.
7. The woman's desire to quit working without giving any reason.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female. Because this research is for pregnant.
Enrollment: 90 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-10 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Number of postpartum women | 6 month
  In the study, R v3.6.1 program was used for Power analysis, alpha error was 5%, beta error was 20%, it was predicted that between the variables as a result of the study process, and a minimum of 90 (45 case groups, 50 control group)

SECONDARY OUTCOMES:
Evaluation of Infant Feeding Attitude | Antenatal and postpartum 6th month
  The Infant Feeding Attitude Scale is used. It includes 17 items with a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Eight statements indicate positive attitude toward breastfeeding and nine statements indicate positive attitude toward formula feeding. The statements indicating positive attitude to breastfeeding were reverse-scored before calculating the total scores of all items. An example for attitude is: "Formula-feeding is more convenient than breastfeeding", and "Breastfeeding increases mother-infant bonding". The total IIFAS score can range from 17 to 85 with higher scores reflecting more positive attitude towards breastfeeding. The total IIFAS is further classified as positive to breastfeeding (a score of 70-85), neutral (a score of 49-69) and positive to formula feeding
Evaluation of Depression Level | Postpartum 7th day, 3rd month, and 6th month
  Edinburgh Postnatal/Postpartum Depression Scale is a self-assessment scale developed to determine the risk of depression in the postpartum period and to measure the level and severity of depression. The scale consists of 10 questions in total. Each question provides a four-point Likert-type measurement. Items in questions 3, 5, 6, 7, 8, 9 and 10 of the scale are scored as 3, 2, 1, 0 and indicate gradually decreasing severity. The items in questions 1, 2 and 4 are scored as 0, 1, 2, 3, indicating increasing severity. The total score of the scale is obtained by summing these items. The minimum total score is 0 and the maximum score is 30. The cut-off score of the scale has been reported as 12/13.
Evaluation of Perception of Insufficient Milk | Postpartum 7th day, 3rd month, and 6th month
  Perception of Insufficient Milk questionnaire is used. The questionnaire consisted of five sections: urine amount, breast condition, stool amount, weight and satisfaction. The characteristics of each section were evaluated on a scale of 0,1,2 points, and a full score of 10 was considered as the best breast milk intake and 7 and below as inadequate breast milk intake.
Evaluation of Breastfeeding Self-Efficacy | Postpartum 7th day, 3rd month, and 6th month
  The Breastfeeding Self-Efficacy Short Form is a 5-point Likert-type scale (1= "I am never sure" and 5 = "I am always sure"). The minimum score is 14 and the maximum score is 70. A higher score indicates higher breastfeeding self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Elif velioğlu, PhDc, Principal Investigator — Marmara University; Nurdan Demirci, Prof, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Kleinpell R, Ely EW, Williams G, Liolios A, Ward N, Tisherman SA. Web-based resources for critical care education. Crit Care Med. 2011 Mar;39(3):541-53. doi: 10.1097/CCM.0b013e318206b5b5. PMID 21169819
- [Result] Maloney S, Haas R, Keating JL, Molloy E, Jolly B, Sims J, Morgan P, Haines T. Breakeven, cost benefit, cost effectiveness, and willingness to pay for web-based versus face-to-face education delivery for health professionals. J Med Internet Res. 2012 Apr 2;14(2):e47. doi: 10.2196/jmir.2040. PMID 22469659
- [Result] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Result] Dennis CL, Faux S. Development and psychometric testing of the Breastfeeding Self-Efficacy Scale. Res Nurs Health. 1999 Oct;22(5):399-409. doi: 10.1002/(sici)1098-240x(199910)22:53.0.co;2-4. PMID 10520192
- [Result] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Derived] Velioglu E, Demirci N. The effect of web-based breastfeeding education given to primiparous pregnant women: a randomised controlled study. Afr J Reprod Health. 2024 Dec 31;28(12):61-72. doi: 10.29063/ajrh2024/v28i12.7. PMID 39764800
- See also: 2018 Turkey Demographic and Health Survey,Hacettepe University Institute of Population Studies Ankara, Turkey — https://fs.hacettepe.edu.tr/hips/dosyalar/Ara%C5%9Ft%C4%B1rmalar%20-%20raporlar/2018%20TNSA/TDHS2018_mainReport_compressed.pdf